CLINICAL TRIAL: NCT03970460
Title: Randomized Clinical Evaluation of Bone Mineral Density Changes Using Two Tibial Base Plate Designs in Primary Total Knee Arthroplasty in Young Patients
Brief Title: Evaluation of Bone Mineral Density Changes Using Two Tibial Base Plate Designs in Primary Total Knee Arthroplasty in Young Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Zimmer Biomet (Industry); CHU de Québec (Unknown)
Responsible Party: Principal Investigator, Michel Malo, Orthopaedic surgeon, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTG-Young
Record Dates: First submitted 2019-05-27; First posted 2019-05-31 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 45-54 y.o / cemented modular metal-backed tibial implant (Active Comparator): This group will undergo a surgery for a knee arthroplasty following standard procedure at our center
  Interventions: Device: Primary TKA with cemented modular metal-backed tibial implant
- 55-59 y.o / cemented modular metal-backed tibial implant (Active Comparator): This group will undergo a surgery for a knee arthroplasty following standard procedure at our center
  Interventions: Device: Primary TKA with cemented modular metal-backed tibial implant
- 45-54 y.o / uncemented Trabecular Metal modular tibial implant (Experimental): This group will undergo a surgery for a knee arthroplasty with a trabecular metal of the tibial implant
  Interventions: Device: Primary TKA with uncemented trabecular metal
- 55-59 y.o / uncemented Trabecular Metal modular tibial implant (Experimental): This group will undergo a surgery for a knee arthroplasty with a trabecular metal of the tibial implant
  Interventions: Device: Primary TKA with uncemented trabecular metal

INTERVENTIONS:
Device: Primary TKA with cemented modular metal-backed tibial implant — Tibial implant will be done with a cemented implant
  Arms: 45-54 y.o / cemented modular metal-backed tibial implant; 55-59 y.o / cemented modular metal-backed tibial implant
Device: Primary TKA with uncemented trabecular metal — Tibial implant will be done with a uncemented implant
  Arms: 45-54 y.o / uncemented Trabecular Metal modular tibial implant; 55-59 y.o / uncemented Trabecular Metal modular tibial implant

SUMMARY:
Arthritic disease in people less than 60 years old is increasingly common. Younger, active individuals often present now to orthopaedic surgeons requiring treatment of knee osteoarthritis. Knee arthroplasty has been offered as a viable option to provide pain relief and improve function in the middle-aged patient.

In a previous study submitted for publication, the investigators have looked at BMD in vivo after total knee replacement comparing two different tibial base plate designs in cemented and uncemented implants in terms of stiffness and modularity, and its effect on bone density changes, synovitis, osteolysis or survivorship. The investigators found a difference of 18% in bone mineral density favoring trabecular metal implant over cemented modular metal-back implant in patient between 55 and 75 years of age. The trabecular metal implant thus behaved as it was expected and preserved bone density in an elderly population.

No randomized clinical trial has looked at cemented titanium tibial insert to uncemented trabecular metal tibia insert in young population. In order to isolate stiffness as study variable, one would aim at randomizing a homogeneous patient population undergoing total knee arthroplasty with implants of similar articular geometry designs with different tibial baseplate, titanium versus trabecular metal. The trabecular metal implant is closer to human bone modulus of elasticity.

DETAILED DESCRIPTION:
THE GOAL OF OUR STUDY IS TO

1. Quantify the amount of bone remodeling 24 months after total knee arthroplasty using sequential dual-energy x-ray absorptiometry of the proximal tibia in younger and more active patients (less than 60 years of age).
2. Evaluate the evolution of functional outcome over a 24 months period using sequential subjective and objective clinical evaluations using the Knee Society Score (KSS) and Knee Injury and Osteoarthritis Outcome Score (KOOS) and Sf-12 v2 in this cohort of patients.
3. There is also an interest in looking at the activity level before and after the surgery (by using the Tegner Activity Level Scale and the UCLA Activity Level Scale) and to determine the ability to return to an active lifestyle and the impact on implant survival.

Two groups will be created:

Group 1: NexGen cemented modular metal-backed tibial implant (Titanium) Group 2: NexGen uncemented Trabecular Metal(TM) modular tibial implant A total of 88 patients will be recruited

ELIGIBILITY:
Inclusion Criteria:

* Tricompartmental osteoarthritis of the knee
* Age, under 60 years old at the time of surgery
* Stable health (the patient should be able to undergo surgery and participate in a follow-up program based upon physical examination and medical history).

Exclusion Criteria:

* Diagnosis of inflammatory joint disease
* Diagnosis of osteonecrosis
* Infection; acute or chronic
* Any current metal hardware on the proximal 25 cm of the tibia
* History, remote or recent, of high tibial osteotomy or tibial plateau fracture
* Any collateral ligamentous instability in the affected knee
* Contra lateral below knee or above knee amputation
* Ongoing Biphosphonate pharmacotherapy
* Presence of clinically significant disease of the cardiovascular, renal, hepatic, hematologic,respiratory, endocrine, neurological, gastrointestinal, genitourinary, immune systems or other medical condition which is not well controlled.
* Participants of a study who have received an investigational drug or device within the last 30 days
* Patients unwilling or unable to cooperate in a follow-up program
* Bone deficit (subchondral cyst)
* Previous contralateral Total Knee Arthroplasty (TKA), ORIF, HTO
* Patella deficiency needing grafting or preventing patella resurfacing

Ages: 45 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-08-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
DEXA Scan | 24 months post-op
  This exam will quantify the amount of bone density at 24 months after total knee arthroplasty. DXA scan can provide accurate, high-quality measurements of periprosthetic bone mineral density (BMD) with minimal precision error and a low coeficient of variation ranging from 1.3% to 4.7%17.
KOOS (knee injury and osteoarthritis outcomes score ) | 2 years post-op
  The Index is self-administered and assesses the 5 subscales: pain (9 questions), other symptoms (7 questions), function in daily living (17 questions), function in sports and recreation (5) and knee related quality of live (4). All subscales are on 100, 100 being the best score, 0 the worst.
  The total score is an average of all subscale
KSS (Knee Society Score) | 2 years post-op
  The original KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.

SECONDARY OUTCOMES:
The 12-item medical outcomes study short form health survey version 2.0 (SF-12v2) | 2 years post-op
  This self-administered generic health status measure is composed of 12 items measuring 3 major health attributes: functional status, well-being, and overall evaluation of health
Lyshom and Tegner | 2 years post-op
  The Lysholm Scale currently consists of eight items that measure: pain (25 points), instability (25 points), locking (15 points), swelling (10 points), limp (5 points), stair climbing (10 points), squatting (5 points), and need for support (5 points). Every question response has been assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions, and may range from 0-100. Higher scores indicate a better outcome with fewer symptoms or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Malo, ND, Principal Investigator — Hôpital Sacré-Coeur de Montréal